CLINICAL TRIAL: NCT06180811
Title: Evaluating the Effectiveness of a Food is Medicine Community Health Worker Program for Pregnant Women: Addressing Social Needs and Improving Health Outcomes
Brief Title: Evaluating the Effectiveness of a Food is Medicine Community Health Worker Program for Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 605512; 90XP0484 (Other Grant/Funding Number: Administration for Children and Families)
Record Dates: First submitted 2023-12-06; First posted 2023-12-26 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pre-Eclampsia; Obesity; Gestational Diabetes; Gestational Hypertension
Keywords: Food is Medicine; Community Health Worker; Social Needs; Medically Tailored Groceries; Randomized Controlled Trial; Maternal and Child Health
MeSH Terms: conditions — Pre-Eclampsia; Obesity; Diabetes, Gestational; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women's Health Delaware Food Farmacy (Experimental): Participants will receive medically tailored groceries (10 meals per person in the household per week from enrollment to 4 weeks after delivery) high in micronutrients that are delivered to their homes weekly. They will also interact weekly with their assigned Community Health Worker to address social needs and patient-centered goals.
  Interventions: Other: Women's Health Delaware Food Farmacy
- Usual Standard of Care (Active Comparator): Participants will receive the usual standard of care.
  Interventions: Other: Usual Standard of Care

INTERVENTIONS:
Other: Women's Health Delaware Food Farmacy — Participants will receive medically tailored groceries (10 meals per person in the household per week from enrollment to 4 weeks after delivery) high in micronutrients that are delivered to their homes weekly. They will also interact weekly with their assigned Community Health Worker to address social needs and patient-centered goals.
  Arms: Women's Health Delaware Food Farmacy
Other: Usual Standard of Care — Participants will receive the usual standard of care.
  Arms: Usual Standard of Care

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial of a food is medicine community health worker intervention called the Women's Health Delaware Food Farmacy compared to the usual standard of care among pregnant ChristianaCare patients at risk for adverse clinical outcomes. The pilot study has three specific aims:

Aim 1: To assess the feasibility of the Women's Health Delaware Food Farmacy and refine the program as needed

Aim 2: To determine the prevalence of and change in social needs

Aim 3: To evaluate the effectiveness of the Women's Health Delaware Food Farmacy on maternal and child health, healthcare utilization, and clinical event outcomes as well as patient-reported outcomes compared to the usual standard of care

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial where eligible pregnant ChristianaCare patients will be identified weekly through an automated list, and patients who consent will be randomized to 1 of 2 arms (Women's Health Delaware Food Farmacy vs. usual standard of care). Participants randomized to the Women's Health Delaware Food Farmacy program arm will receive medically tailored groceries that are high in micronutrients critical for a healthy pregnancy. The food provided will be the equivalent of 10 meals per person in the household per week and will be delivered to participants weekly from enrollment to 4 weeks after giving birth. Participants will receive culinary equipment and training, recipes, and educational nutrition videos and will interact weekly with their assigned Community Health Worker to address social needs and patient-centered goals. Participants randomized to the usual standard of care arm will continue to receive their standard of care management.

All participants will complete a questionnaire with patient-reported outcomes (i.e., food insecurity, dietary intake, health-related quality of life, and cost-related medication underuse) at baseline and postpartum and a patient experience survey postpartum related to their experiences receiving prenatal care and giving birth at ChristianaCare. In addition, maternal and child health, healthcare utilization, and clinical event outcomes will be documented for all participants via electronic health records and assessed retrospectively. Quantitative indicators related to feasibility (i.e., acceptability, demand, and implementation) will be collected such as program satisfaction, program enrollment and retention, meals provided to participants and their household, food consumption, and interactions with assigned Community Health Worker.

Aim 1: To assess the feasibility of the Women's Health Delaware Food Farmacy and refine the program as needed

H1. Primary outcomes. The investigators hypothesize that the Women's Health Delaware Food Farmacy will: (a) prove acceptable to participants, as measured by program satisfaction; (b) meet demand, as measured by project recruitment and retention, number of meals provided to participants and their household, and number of people providing food for; and (c) prove implementable, as measured by food consumption, number of Community Health Worker interactions, number of educational videos watched, number of recipes reviewed, and number of meal preparation sessions.

Aim 2: To determine the prevalence of and change in social needs

H2. Primary outcome. Social needs will be identified by administering the ChristianaCare Social Determinants of Health Screener and resource referrals will be sent on participants' behalf to support their social needs, both of which are the usual standard of care. The investigators hypothesize that social needs will be identified through the ChristianaCare Social Determinants of Health Screener, and that compared to baseline, participants at postpartum will experience reductions in their social needs. The investigators also hypothesize there will be some participants whose social needs will not be resolved due to a lack of community resources.

Aim 3: To evaluate the effectiveness of the Women's Health Delaware Food Farmacy on maternal and child health, healthcare utilization, and clinical event outcomes as well as patient-reported outcomes compared to the usual standard of care

H3a. Primary outcomes. Maternal and child health outcomes: The investigators hypothesize that compared to usual standard of care, the Women's Health Delaware Food Farmacy group will demonstrate improvements in maternal and child health outcomes (e.g., preeclampsia and small for gestational age) from baseline to postpartum.

H3b. Primary outcomes. Maternal and child healthcare utilization outcomes: The investigators hypothesize that compared to usual standard of care, the Women's Health Delaware Food Farmacy group will demonstrate reductions in maternal and child healthcare utilization outcomes (e.g., neonatal intensive care unit [NICU] admission and maternal length of stay) from baseline to postpartum.

H3c. Primary outcomes. Maternal and child clinical event outcomes: The investigators hypothesize that compared to usual standard of care, the Women's Health Delaware Food Farmacy group will demonstrate reductions in maternal and child clinical event outcomes (e.g., cesarean delivery and fetal death) from baseline to postpartum.

H3d. Secondary outcomes. Patient-reported outcomes: The investigators hypothesize that compared to usual standard of care, the Women's Health Delaware Food Farmacy group will demonstrate improvements in patient-reported outcomes (i.e., food insecurity, dietary intake, health-related quality of life, and cost-related medication underuse) from baseline to postpartum.

ELIGIBILITY:
Inclusion Criteria:

* ChristianaCare Women's Health patient
* 18 years or older
* 4 to 14 weeks pregnant
* Singleton pregnancy
* Medicaid
* BMI of 30 or higher
* Reside in New Castle County

Exclusion Criteria:

* Current diagnosis of type 1 or type 2 diabetes
* Multiple pregnancy
* Currently enrolled in another Community Health Worker program
* Not able to store and prepare meals
* Diagnosed with severe medical comorbidities that might interfere with their ability to participate in the intervention, such as severe psychiatric illness or imminent hospitalization
* Not able to understand and communicate effectively in English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Social Determinants of Health | Changes from baseline to 2-6 weeks after delivery
  Measured with ChristianaCare Social Determinants of Health Screener; Number of socials needs range from 0-11, higher scores indicate greater number of social needs
Gestational Weight Gain | Changes from baseline to 2-6 weeks after delivery
  Observed gestational weight gained
Body Mass Index | Changes from baseline to 2-6 weeks after delivery
  Observed body mass index changes
Gestational Diabetes | From baseline to delivery
  Occurrence of gestational diabetes
Gestational Hypertension | From baseline to delivery
  Occurrence of gestational hypertension
Systolic and Diastolic Blood Pressure | Changes from baseline to 2-6 weeks after delivery
  Observed systolic and diastolic blood pressure
Preeclampsia | From baseline to 2-6 weeks after delivery
  Occurrence of preeclampsia and week diagnosed during pregnancy
Hydramnios | From baseline to delivery
  Occurrence of hydramnios
Gestational Age | At delivery
  Baby's gestational age at birth
Small for Gestational Age | At delivery
  Birth weight less than 10th percentile based on gestational age
Preterm Birth | At delivery
  Preterm birth less than 37 weeks
Fetal Macrosomia | At delivery
  Birth weight greater than 90th percentile based on gestational age
Cesarean Delivery | At delivery
  Occurrence of cesarean delivery including those planned and unplanned
Fetal Death | From baseline to delivery
  Occurrence of fetal death
NICU Admission | Within 48 hours after delivery
  Occurrence of NICU admission for any reason
NICU Length of Stay | From NICU admission date to NICU discharge date, assessed up to 90 days
  Number of days baby was admitted to NICU
Maternal Length of Stay | From delivery date to hospital discharge date, assessed up to 90 days
  Number of days hospitalized following delivery
Postpartum Admission | From delivery discharge to 90 days after
  Number of postpartum hospital admissions for any reason
Postpartum Admission Length of Stay | From postpartum admission date to hospital discharge date, assessed up to 90 days
  Number of days hospitalized
Hospital Admission | From baseline up to delivery
  Number of hospital admissions for any reason
Hospital Admission Length of Stay | From admission date to hospital discharge date, assessed up to 90 days
  Number of days hospitalized
Emergency Room Visit | From baseline to 90 days after delivery
  Number of emergency room visits for any reason

SECONDARY OUTCOMES:
Food Insecurity | Changes from baseline to 2-6 weeks after delivery
  Measured with United States Department of Agriculture Household Food Security Survey Module 6-Item Short Form, 30-day; Scores range from 0-6, higher scores indicate lower food security
Dietary Intake | Changes from baseline to 2-6 weeks after delivery
  Measured with Dietary Screener Questionnaire (DSQ-10) and six items from Dietary Screener Questionnaire (DSQ-26); Scores will be calculated using the National Cancer Institute's scoring algorithms
Health-Related Quality of Life | Changes from baseline to 2-6 weeks after delivery
  Measured with Centers for Disease Control and Prevention's Health-Related Quality of Life (HRQOL-4) scale; Number of healthy days range from 0-30, higher scores indicate greater number of healthy days
Cost-Related Medication Underuse | Changes from baseline to 2-6 weeks after delivery
  Measured with Cost-Related Medication Underuse; Scores range from 0-4, scores greater than 0 indicate cost-related medication underuse

CONTACTS AND LOCATIONS:
Locations (1):
- ChristianaCare Christiana Hospital, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT06180811/SAP_000.pdf